CLINICAL TRIAL: NCT06867094
Title: A Phase 2, Multinational, Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study to Evaluate the Efficacy and Safety of SAR441566 in Adults With Moderate-to-severe Ulcerative Colitis
Brief Title: A Study to Investigate Efficacy and Safety of SAR441566 in Patients With Ulcerative Colitis
Acronym: SPECIFI-UC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRI17822; U1111-1308-9729 (Other: WHO); 2025-520705-12 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Colitis Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SAR441566 dose regimen 1 (Experimental): Participants will receive SAR441566 dose regimen 1
  Interventions: Drug: SAR441566
- SAR441566 dose regimen 2 (Experimental): Participants will receive SAR441566 dose regimen 2
  Interventions: Drug: SAR441566
- SAR441566 dose regimen 3 (Experimental): Participants will receive SAR441566 dose regimen 3
  Interventions: Drug: SAR441566
- Placebo (Placebo Comparator): Participants will receive SAR441566-matching placebo
  Interventions: Drug: SAR441566 matching Placebo

INTERVENTIONS:
Drug: SAR441566 — Pharmaceutical form: Tablet Route of administration: Oral
  Arms: SAR441566 dose regimen 1; SAR441566 dose regimen 2; SAR441566 dose regimen 3
Drug: SAR441566 matching Placebo — Pharmaceutical form: Tablet Route of administration: Oral
  Arms: Placebo

SUMMARY:
This is a Phase 2, multinational, multicenter, randomized, double-blind, placebo-controlled, dose ranging study to evaluate the efficacy and safety of SAR441566 in adults with moderate-to-severe UC. The primary objective of this study is to assess efficacy of different doses of SAR441566 on clinical remission in participants with moderate-to-severe ulcerative colitis.

This study will include a screening period of up to 28 days (+ 7 calendar days if needed) followed by the main study treatment period of 52 weeks which will be comprised of a double blind (DB) treatment period with 12 weeks of induction period followed by a maintenance period of 40 weeks and 2-week follow-up after end of treatment.

Additionally, an Open Label (OL) period of up to 40 weeks will be offered to eligible participants.

* The study duration will be up to 59 weeks.
* The treatment duration will be up to 52 weeks in the DB arm and up to 40 weeks in the OL arm.
* The number of visits will be 12 for the main study treatment period and 8 for the OL treatment period.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* Male or female participants aged 18 to 75 years inclusive, at the time of signing the informed consent
* Participants who have clinical evidence of active UC for ≥3 months before screening and confirmed by endoscopy during the screening period
* Active moderate-to-severe UC at screening as defined by a modified Mayo Score (mMS) of 5 to 9 (without the Physician global Assessment (PGA), with a minimum rectal bleeding (RB) subscore ≥1, a minimum stool frequency (SF) subscore ≥1, a mMES ≥2 confirmed by central reader, a minimum sum of all subscores of 5, and a disease extent >15 cm from the anal verge
* Must have received prior treatment for UC (either "a" or "b" below or combination of both):

  1. No prior exposure to Advanced Therapy (AT), but having inadequate response to, loss of response to or intolerance to standard treatment with any of the following compounds: 5-ASA, 6-MP, AZA, MTX, oral or intravenous (IV) corticosteroids or history of corticosteroid dependence (defined an inability to successfully taper corticosteroids without recurrence of UC) OR
  2. Inadequate response to, loss of response to or intolerance to treatment with ≥1 approved AT such as a biologic agent (such as TNF antagonists, anti-integrin other than natalizumab, anti-IL-12/23, anti-IL-23, or experimental biologic UC therapeutics), or a small molecule (such as a JAKi or S1PRm) for UC
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Participants with active CD, indeterminate colitis, ischemic colitis, microscopic colitis
* Participants with the following ongoing known complications of UC: fulminant colitis, toxic megacolon, or any other manifestation that might require bowel surgery while enrolled in the study
* Participant with prior colectomy, ostomy or ileoanal pouch, or anticipated colectomy during their participation in the study
* Participants with fecal sample positive for ova or parasites, bacterial pathogens, or positive for Clostridium difficile B toxin in stools
* Participants with active tuberculosis (TB) or a history of incompletely treated active TB or latent TB infection per local guidelines
* Participants with Positive Hepatitis B surface antigen (HBsAg), or Hepatitis B core antibody (HBcAb) and/or Hepatitis C virus antibody (HCVAb) at the screening visit
* Participants with any other active, chronic or recurrent infection, including recurrent or disseminated herpes zoster or disseminated herpes simplex
* Participants with a known history of human immunodeficiency virus (HIV) infection or positive HIV-1 or HIV-2 serology at screening
* Participants presenting with active malignancies, lymphoproliferative disease, or recurrence of either, within the 5 years before screening
* If the participant has extensive colitis for ≥8 years or disease limited to left side of colon (ie, distal to splenic flexure) for >10 years, regardless of age, a colonoscopy within 1 year of the screening visit is required to survey for dysplasia. Participants with dysplasia or cancer identified on biopsies will be excluded.
* Female participants who is pregnant, breastfeeding, or is considering becoming pregnant during the study or within 3 months after the last dose of study drug
* Infection(s) requiring treatment with IV anti-infectives within 30 days prior to the screening visit or oral/intramuscular anti-infectives within 14 days prior to the screening visit
* Participants requiring or receiving any parental nutrition and/or exclusive enteral nutrition
* Participants who received cyclosporine, tacrolimus, mycophenolate mofetil, or thalidomide within 30 days prior to screening
* Participants who received fecal microbial transplantation within 30 days prior to screening
* Participants who have ever been exposed to natalizumab (Tysabri®) or oral carotegrast methyl (Carogra®)
* Participants who received IV corticosteroids within 14 days prior to screening or during screening period
* Screening laboratory and other analyses show abnormal results.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2027-07-29 (Estimated); Study Completion 2028-05-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving clinical remission at Week 12 by modified Mayo Score (mMS) | Week 12
  Clinical remission by modified Mayo score (mMS) is defined as a mMS ≤2 with no subscore >1 (stool frequency [SF] of 0 or 1 with at least a 1-point decrease from baseline, rectal bleeding [RB] of 0 and modified Mayo Endoscopic Subscore [mMES] of 0 or 1 where 1 does not include friability).
  Each component of the mMS (SF, RB, and mMES) is scored from 0 to 3. The total mMS ranges from 0 to 9 with higher scores indicating greater disease severity.

SECONDARY OUTCOMES:
Proportion of participants achieving clinical response at Week 12 by modified Mayo Score (mMS) | Week 12
  Clinical response by modified Mayo score (mMS) is defined as a decrease from baseline in the mMS of ≥2 points and an improvement of ≥30% from baseline plus a decrease in rectal bleeding (RB) subscore ≥1 or an absolute RB subscore ≤1.
  Each component of the mMS (SF, RB, and mMES) is scored from 0 to 3. The total mMS ranges from 0 to 9 with higher scores indicating greater disease severity.
Proportion of participants achieving clinical response at Week 12 by full Mayo score (MS) | Week 12
  Clinical response by full Mayo score (MS) is defined as a decrease from baseline in the MS of ≥3 points and an improvement of ≥30% from baseline plus a decrease in rectal bleeding (RB) subscore ≥1 or an absolute RB subscore ≤1.
  The MS (also referred to as the full Mayo Score) is a composite index designed to measure ulcerative colitis (UC) disease activity and consists of 4 subscores: RB and SF, which are patient-reported subscores, Physician's global assessment (PGA), and endoscopic findings. Individual items are rated 0 to 3, giving the composite score a maximum of 12, with higher scores indicating greater disease severity.
Proportion of participants achieving clinical remission at Week 12 by full Mayo score (MS) | Week 12
  Clinical remission by full Mayo score (MS) is defined as a MS ≤2 with no score >1.
Proportion of participants achieving the combination of patient-reported outcome 2 (PRO2) remission and endoscopic remission at Week 12 | Week 12
  Patient-reported outcome 2 (PRO2) remission is defined as PRO2 score ≤1 with rectal bleeding (RB) of 0, and endoscopic remission is defined as mMES of 0.
  PRO2 score is defined as the sum of Mayo SF and RB subscores.
Proportion of participants achieving endoscopic remission at Week 12 | Week 12
  Endoscopic remission is defined as mMES=0.
Change from baseline in PRO2 from randomization to Week 12 | From Baseline to Week 12
  PRO2 score is defined as the sum of the Mayo SF and RB subscores.
Proportion of participants achieving endoscopic response at Week 12 | Week 12
  Endoscopic response is defined as mMES decrease of at least 1 point.
Proportion of participants achieving endoscopic improvement at Week 12 | Week 12
  Endoscopic improvement is defined as mMES of 0 or 1 where 1 does not include friability.
Proportion of participants achieving HEMI at Week 12 | Week 12
  Histologic endoscopic mucosal improvement (HEMI) is defined by achievement of modified Mayo endoscopic improvement (mMES of 0 or 1 where 1 does not include friability) and histological improvement (original Geboes Score [OGS] ≤3.1).
Plasma predose concentrations of SAR441566 at selected visits | Up to Week 52
Plasma postdose concentrations of SAR441566 at selected visits | Up to Week 52
Number of participants with any treatment-emergent adverse events (TEAEs) during induction and maintenance treatment period | Up to Week 52
Number of participants with any treatment-emergent adverse events (TEAEs) during open-label treatment period | From Week 12 to Week 52
Proportion achieving Inflammatory Bowel Disease Questionnaire (IBDQ) remission at Week 12 | Week 12
  Inflammatory Bowel Disease Questionnaire (IBDQ) remission is considered as an IBDQ-32 total score ≥170 points.
  IBDQ is designed to capture the patient's experience of IBD on 4 domains of functioning and well-being: bowel and systemic symptoms and emotional and social function. The total IBDQ score ranges from 32 to 224 which indicates better quality of life.
Proportion of participants achieving Inflammatory Bowel Disease Questionnaire (IBDQ) response at Week 12 | Week 12
  Inflammatory Bowel Disease Questionnaire (IBDQ) response is defined as an increase from baseline in the total IBDQ score in the range of 16 to 32 points.

CONTACTS AND LOCATIONS:
Locations (105):
- United States (18):
  - GI Alliance - Arizona Digestive Health - Sun City- Site Number : 8400003, Sun City, Arizona
  - Bristol Hospital- Site Number : 8400017, Bristol, Connecticut
  - Novum Research- Site Number : 8400018, Clermont, Florida
  - Clinical Research of Osceola- Site Number : 8400012, Kissimmee, Florida
  - Wellness Clinical Research - Miami Lakes - 8181 Northwest 154th Street- Site Number : 8400002, Miami Lakes, Florida
  - GCP Clinical Research- Site Number : 8400016, Tampa, Florida
  - GI Alliance - Glenview- Site Number : 8400005, Glenview, Illinois
  - Illinois Gastroenterology Group- Site Number : 8400004, Gurnee, Illinois
  - University of Michigan Health System - Ann Arbor- Site Number : 8400010, Ann Arbor, Michigan
  - Icahn School of Medicine at Mount Sinai- Site Number : 8400001, New York, New York
  - Queens Village Primary Medical Center- Site Number : 8400011, Queens Village, New York
  - NexGen Research- Site Number : 8400020, Lima, Ohio
  - Frontier Clinical Research - Uniontown- Site Number : 8400006, Uniontown, Pennsylvania
  - Gastro Health & Nutrition- Site Number : 8400007, Katy, Texas
  - SI Research Associates- Site Number : 8400019, Lubbock, Texas
  - Texas Digestive Disease Consultants - Southlake- Site Number : 8400015, Southlake, Texas
  - University of Washington Medical Center- Site Number : 8400014, Seattle, Washington
  - Washington Gastroenterology - Tacoma- Site Number : 8400009, Tacoma, Washington
- Argentina (5):
  - Investigational Site Number : 0320004, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number : 0320003, Buenos Aires
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320005, Buenos Aires
- Investigational Site Number : 0360003, Kurralta Park, South Australia, Australia
- Austria (3):
  - Investigational Site Number : 0400003, Graz
  - Investigational Site Number : 0400002, Salzburg
  - Investigational Site Number : 0400001, Vienna
- Belgium (2):
  - Investigational Site Number : 0560002, Ghent
  - Investigational Site Number : 0560001, Leuven
- Brazil (2):
  - Hospital de Clinicas de Porto Alegre- Site Number : 0760002, Porto Alegre, Rio Grande do Sul
  - Hospital Ernesto Dornelles- Site Number : 0760003, Porto Alegre, Rio Grande do Sul
- Bulgaria (3):
  - Investigational Site Number : 1000001, Burgas
  - Investigational Site Number : 1000003, Rousse
  - Investigational Site Number : 1000002, Sofia
- Canada (3):
  - Investigational Site Number : 1240004, Kentville, Nova Scotia
  - Investigational Site Number : 1240005, Richmond Hill, Ontario
  - Investigational Site Number : 1240001, Québec, Quebec
- Chile (3):
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
- China (9):
  - Investigational Site Number : 1560002, Guangzhou
  - Investigational Site Number : 1560001, Hangzhou
  - Investigational Site Number : 1560003, Huizhou
  - Investigational Site Number : 1560004, Jiazhuang
  - Investigational Site Number : 1560014, Linhai
  - Investigational Site Number : 1560008, Luoyang
  - Investigational Site Number : 1560005, Shanghai
  - Investigational Site Number : 1560007, Shanghai
  - Investigational Site Number : 1560011, Wuhan
- Czechia (2):
  - Investigational Site Number : 2030001, Olomouc
  - Investigational Site Number : 2030002, Ostrava
- France (3):
  - Investigational Site Number : 2500003, Nice
  - Investigational Site Number : 2500001, Toulouse
  - Investigational Site Number : 2500002, Vandœuvre-lès-Nancy
- Georgia (3):
  - Investigational Site Number : 2680002, Tbilisi
  - Investigational Site Number : 2680003, Tbilisi
  - Investigational Site Number : 2680001, Tbilisi
- Germany (7):
  - Investigational Site Number : 2760005, Berlin
  - Investigational Site Number : 2760008, Berlin
  - Investigational Site Number : 2760010, Duisburg
  - Investigational Site Number : 2760009, Frankfurt
  - Investigational Site Number : 2760003, Hanover
  - Investigational Site Number : 2760011, Tübingen
  - Investigational Site Number : 2760006, Ulm
- Greece (3):
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000003, Athens
  - Investigational Site Number : 3000002, Heraklion
- India (7):
  - Investigational Site Number : 3560005, Hyderabad
  - Investigational Site Number : 3560003, Jaipur
  - Investigational Site Number : 3560009, Jaipur
  - Investigational Site Number : 3560002, Kolkata
  - Investigational Site Number : 3560007, Secunderabad
  - Investigational Site Number : 3560001, Surat
  - Investigational Site Number : 3560010, Visakhapatnam
- Italy (9):
  - Investigational Site Number : 3800006, Genoa, Genova
  - Investigational Site Number : 3800002, Milan, Milano
  - Investigational Site Number : 3800003, Rozzano, Milano
  - Investigational Site Number : 3800008, Naples, Napoli
  - Investigational Site Number : 3800001, Padua, Padova
  - Investigational Site Number : 3800010, Turin, Torino
  - Investigational Site Number : 3800007, Alessandria
  - Investigational Site Number : 3800009, Palermo
  - Investigational Site Number : 3800004, Pisa
- Japan (14):
  - Investigational Site Number : 3920005, Kashiwa, Chiba
  - Investigational Site Number : 3920014, Kure, Hiroshima
  - Investigational Site Number : 3920003, Sapporo, Hokkaido
  - Investigational Site Number : 3920007, Sapporo, Hokkaido
  - Investigational Site Number : 3920009, Morioka, Iwate
  - Investigational Site Number : 3920013, Yokohama, Kanagawa
  - Investigational Site Number : 3920002, Bunkyo, Tokyo
  - Investigational Site Number : 3920011, Kodaira, Tokyo
  - Investigational Site Number : 3920015, Minato-ku, Tokyo
  - Investigational Site Number : 3920006, Kofu, Yamanashi
  - Investigational Site Number : 3920012, Hiroshima
  - Investigational Site Number : 3920016, Kagoshima
  - Investigational Site Number : 3920001, Niigata
  - Investigational Site Number : 3920010, Osaka
- Poland (5):
  - Investigational Site Number : 6160008, Oświęcim, Lesser Poland Voivodeship
  - Investigational Site Number : 6160005, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6160004, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160001, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160002, Rzeszów, Podkarpackie Voivodeship
- Turkey (Türkiye) (3):
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7920003, Izmir
  - Investigational Site Number : 7920001, Mersin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: DRI17822 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26594&tenant=MT_SNY_9011